CLINICAL TRIAL: NCT05966740
Title: Safety and Effectiveness of Pradaxa Oral Pellet Formulation for Treatment of Acute Venous Thromboembolic Events (VTE) and/or for Risk Reduction of Recurrence of VTE in Pediatric Patients Aged 3 Months to Less Than 12 Years in a Real World Setting: a Prospective Non-interventional Study Conducted in the United States
Brief Title: A Study in the United Sates That Looks at the Safety and Effectiveness of Pradaxa Pellets in Children Aged 3 Months to Less Than 12 Years Who Need Treatment of a Blood Clot or Who Have Had a Blood Clot and Are at Risk of Developing Another Blood Clot
Status: Terminated | Type: Observational
Why Stopped: Low study enrolment.
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Children's Hospital Acquired Thrombosis consortium (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1160-0309
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients with VTE and/or at risk for VTE

SUMMARY:
The main research question of this study is to obtain further safety and effectiveness data on Pradaxa Pellets in children aged 3 months to less than 12 years in routine clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients aged 3 months to less than 12 years at the time of Pradaxa Pellets initiation

* Written informed consent from parents/care givers and patient assent if age appropriate
* Initiation of Pradaxa Pellets administration either as initial or subsequent therapy:

  * Treatment of VTE
  * Treatment to reduce the risk of recurrence of VTE

Exclusion Criteria:

* Participation in any randomized clinical trial or use of investigational product, participation in any other observational study is not an exclusion
* Any contraindications to Pradaxa Pellets according to the US Prescribing Information.
* Previous participation in this study.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged 3 months to less than 12 years, who may be considered for anticoagulation with Pradaxa Pellets due to venous thromboembolic events (VTE), are usually treated in neonatology, pediatric general surgery, cardiac surgery or intensive care units. Pediatric patients with anticoagulation with Pradaxa Pellets for the prevention of recurrent VTE are usually evaluated by pediatric hematologists in pediatric hematology units. Any of these patients that are prescribed Pradaxa pellets may be considered for inclusion into this study.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of clinically relevant bleeding events | Up to week 52

SECONDARY OUTCOMES:
Occurrence of recurrent Venous Thromboembolic Event (VTE) | Up to week 52
Mortality related to thrombotic or thromboembolic events | Up to week 52
Occurence of all bleeding events | Up to week 52
Occurrence of post-thrombotic syndrome (PTS) | Up to week 52
Incidence of adverse events (AEs) | Up to week 52
Incidence of serious adverse events (SAEs) | Up to week 52
Thrombotic burden at the end of the treatment period vs baseline, i.e. image-based resolution status of the thrombus (complete response, partial response, stable disease, progressive disease) | Baseline and up to week 12
Recurrence of VTE while on treatment | Up to week 52
Duration of treatment with dabigatran etexilate | Up to week 52
Compliance with dabigatran etexilate treatment | Up to week 52

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of California, San Diego, La Jolla, California
  - Rady Children's Hospital, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Indiana Hemophilia & Thrombrosis Center, Indianapolis, Indiana
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - MUSC (Medical university of South Carolina), Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Dell Children's Ascension, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com